CLINICAL TRIAL: NCT03582839
Title: Effects of an Internet Use Disorder and Internet Gaming Disorder Early Intervention Program
Acronym: PROTECT+
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pädagogische Hochschule Heidelberg (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Principal Investigator, Dr. Katajun Lindenberg, Jun.-Prof. Dr. K. Lindenberg, Pädagogische Hochschule Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH Heidelberg
Record Dates: First submitted 2018-06-04; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PROTECT+ (Experimental): The PROTECT+ intervention group is a self-selected sample, which receives the PROTECT+ group therapy (4 modules in 4 subsequent weeks à 100 min). Participants are assessed at T1 (baseline), T2 (post treatment, 1-month follow-up), T3 (4-months follow-up), and T4 (12-months follow-up).
  Interventions: Behavioral: PROTECT+

INTERVENTIONS:
Behavioral: PROTECT+ — The early intervention PROTECT+ consists of a cognitive-behavioral 4-session brief-protocol (100 minutes) and targets empirically identified risk factors of (I)GD/IUD, i.e. (1) boredom and motivational problems, (2) procrastination and performance anxiety, (3) social behavior and (4) emotion regulation. It addresses both risk-reduction and strength-promotion by cognitive behavioral (CB) interventions such as (1) psychoeducation, (2) cognitive restructuring (identification and modification of dysfunctional cognition), (3) behavior modification (improving problem solving skills, training of functional behavior and reinforcement) as well as (4) improving emotion regulation (training of sensory, imaginative and mindfulness based techniques).

SUMMARY:
Background. In the last two decades Internet usage has grown vastly. Pathological Internet usage (IUD; Internet Use Disorder) is associated with severe mental health problems affecting social, academic and daily life functioning. Internet Gaming Disorder (IGD) has been already included in the DSM-V. Recently, the WHO declared to include Gaming Disorder (GD) in the upcoming ICD-11. Despite the increasing rates of adolescents with IUD and (I)GD, affected people are treated unsystematically and there is a lack of evidence based treatment programs. PROTECT+ is a low-threshold, cognitive behavioral short-term group intervention.

Methods. 54 patients, aged 9-19 years, received PROTECT+ intervention in Heidelberg, Germany. The PROTECT+ intervention group underwent a cognitive-behavioral 4-session group therapy. Follow-up data were collected at 1, 4, and 12 months after admission. Primary outcome was the change in (I)GD and IUD related symptoms at the 12-months follow-up. Secondary outcomes were changes in comorbid symptoms as well as in problem solving, cognitive restructuring and emotion regulation skills

Discussion. Treatment of IUD and IGD is still in its early stages. Recent reviews report increasing research on treatment but also a lack of well-designed studies and evidence based treatment programs. The PROTECT+ intervention is a theory driven and evidence based therapy program which is based on the PROTECT preventive intervention in school settings. In the intervention group a reduction of (I)GD and IUD symptom severity is expected over 12 months.

ELIGIBILITY:
Inclusion Criteria:

Adolescents aged 9 to 19 years Self-selection

Exclusion Criteria:

Severe comorbid mental health disorder

Ages: 9 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2018-12-23 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Changes in IUD symptom severity (self-report) | baseline, 1 month, 4-months, 12-months
  IUD symptom severity is assessed by the Compulsive Internet Use Scale (CIUS; Meerkerk, Van Den Eijnden, Vermulst & Garretsen, 2009). The CIUS is a broadly used and validated questionnaire including 14 Items assessing IUD.
Changes in (I)GD/IUD symptom severity (self-report and parental report) | baseline, 1 month, 4-months, 12-months
  (I)GD/IUD symptom severity is assessed via self-reports and via parental reports by the Video Game Dependency Scale (Computerspielabhängigkeitsskala; CSAS; Rehbein, Baier, Kleimann & Mößle, 2015). The CSAS questionnaire has been adapted by including non-gaming IU.
Changes in (I)GD/IUD symptom severity (Clinical Interview based on DSM-5) | 12-months
  At 12-months follow-up, we conduct a clinical interview based on the criteria of IGD according to the DSM-5. We adapted the criteria by non-gaming subtypes to assess IUD.

SECONDARY OUTCOMES:
Emotion Regulation | baseline, 1 month, 4-months, 12-months
  For the measurement of emotion regulation the German Questionnaire for Assessment of Emotion Regulation in Children and Adolescents (Fragebogen zur Erhebung der Emotionsregulation bei Kindern und Jugendlichen; FEEL-KJ; Grob & Smolenski, 2011) is used. The questionnaire includes a measure of functional and dysfunctional emotion regulation strategies for the negative emotions fear, sadness and anger.
Depressive Symptoms | baseline, 1 month, 4-months, 12-months
  Depressive symptoms are assessed using the German Depression Inventory for Children and Adolescents (Depressionsinventar für Kinder und Jugendliche; DIKJ; Stiensmeier-Pelster, Braune-Krickau, Schürmann & Duda, 2014; Stiensmeier-Pelster, Schürmann & Duda, 1989). The instrument allows for the detection and estimation of severity of depressive disorders according to the DSM-5 criteria (American Psychiatric Association, 2013).
Comorbid emotional, oppositional, antisocial and attention deficit/ hyperactivity disorders | baseline, 1 month, 4-months, 12-months
  Comorbid Psychopathology is assessed using the Strength and Difficulties Questionnaire (SDQ; Goodman, Meltzer & Bailey, 2003).
  It includes the 5 scales (1) emotional problems, (2) behavior problems, (3) hyperactivity/ attention deficits, (4) interpersonal problems with peers and (5) prosocial behavior and can be used for epidemiological research and as an indicator for emotional, oppositional, antisocial and attention deficit/ hyperactivity disorder. The Total Difficulties Score of the SDQ indicates the risk for developing a mental health disorder.
Anxiety Disorders: Social Anxiety | baseline, 1 month, 4-months, 12-months
  We assess social anxiety using the German version of the Social Interaction Anxiety Scale (SIAS; Mattick & Clarke, 1998; Stangier, Heidenreich, Berardi, Golbs & Hoyer, 1999). This questionnaire assesses anxiety in social interactions and allows for detection and the estimation of severity of social anxiety disorders.
Anxiety Disorders: Performance and School Anxiety | baseline, 1 month, 4-months, 12-months
  We assess performance and school anxiety with the 7th scale of the German adaption of the Fear Survey Schedule for Children - Revised (Phobiefragebogen für Kinder und Jugendliche; PHOKI Döpfner, Schnabel, Goletz & Ollendick, 2006; Muris & Ollendick, 2002).
Procrastination | baseline, 1 month, 4-months, 12-months
  Procrastination is assessed with the German Questionnaire for Procrastination (Allgemeiner Prokrastinationsfragebogen; APROF; Höcker, Engberding & Rist, 2013).
Social Behavior and Learning Behavior | baseline, 1 month, 4-months, 12-months
  For ratings of social competent behavior and academic motivation, we use the German Student Assessment List for Social and Learning Behavior (Schülereinschätzliste für Sozial- und Lernverhalten; SSL; Petermann & Petermann, 2014; Petermann, Petermann & Lohbeck, 2014).
Self-Efficacy | baseline, 1 month, 4-months, 12-months
  Self- efficacy is rated on the German Self-Efficacy Scale (Skala zu Allgemeinen Selbstwirksamkeitserwartung; SWE; Schwarzer & Jerusalem, 1999).

CONTACTS AND LOCATIONS:
Overall Officials: Katajun Lindenberg, PhD, Principal Investigator — Institut für Psychologie der Pädagogischen Hochschule Heidelberg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Szasz-Janocha C, Vonderlin E, Lindenberg K. Treatment outcomes of a CBT-based group intervention for adolescents with Internet use disorders. J Behav Addict. 2020 Nov 16;9(4):978-989. doi: 10.1556/2006.2020.00089. PMID 33216013